CLINICAL TRIAL: NCT05754801
Title: Yunzhi Essence to Improve the Quality of Life of Patients With Advanced Stage of Cancer: A Randomized, Double-blinded, Placebo-controlled Trial
Brief Title: Yunzhi Essence to Improve the Quality of Life of Patients With Advanced Stage of Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Lin Zhixiu, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Yunzhi study
Record Dates: First submitted 2022-12-28; First posted 2023-03-06 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Cancer; Palliative Care
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active treatment (Yunzhi Essence) (Experimental): Subjects will take 2 Yunzhi capsules, 4 times daily, for 6 months.
  Interventions: Drug: Yunzhi Essence
- Placebo (Placebo Comparator): Subjects will take 2 placebo capsules, 4 times daily, for 6 months
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Yunzhi Essence — Yunzhi Essence capsule
  Other Names: Yunzhi
  Arms: Active treatment (Yunzhi Essence)
Other: Placebo — Placebo capsules
  Arms: Placebo

SUMMARY:
A randomized, double-blinded, placebo-controlled clinical trial using a Chinese Medicine 'Coriolus Versicolor for improving the quality of life of patients with advanced-stage cancer. Subjects will be randomized into a treatment group or placebo group for 6 months.

DETAILED DESCRIPTION:
According to the Compendium of Materia Medica, a classic encyclopedia for Chinese medicines written by the venerated Physician Li ShiZhen of the Ming dynasty, Yunzhi (Coriolus Versicolor) is treasured as a superbly valuable herb as it not only can strengthen and consolidate the body's resistance, as well as reinforce and nourish a person's marrow and kidney essence and also is harmless to patients. Recent research found that the extract from Yunzhi, named as polysaccharide-peptide (PSP), could inhibit the growth of human hematoma cell line & sarcoma and was proved to have direct anti-cancer effects.

Quality of life (QOL) of patients is the ultimate goal of palliative care as endorsed by the World Health Organization (WHO) in 1990. When survival is limited in advanced incurable diseases, quality of life is most important. Patients with advanced cancer (palliative) often manifest numerous physical and psychological symptoms and a poor quality of life. While maintenance of the quality of life of advanced cancer patients is important, the physical dimension of quality of life still needs improvement, especially in the palliative stage. To date, there is no specific supportive Traditional Chinese Medicine(TCM)-related products that have been proven in randomized controlled trials for alleviating these debilitating symptoms and improving their quality of life. The present study aims to scientifically evaluate whether a Yunzhi product named G.E. Yunzhi-Essence is effective and safe in improving the QOL of palliative patients with advanced cancer.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with advanced cancer according to the definition from American Cancer Society;
* According to the experience of the doctor, by using Palliative Prognostic Index (score>4), integrated with past cases and professional knowledge judged to have life expectancy not less than six months to two years;
* Abbreviated mental test (AMT) score of 6 or above;
* Voluntarily participate in this clinical trial and sign the informed consent form (acceptance of close relatives signed informed consent on behalf of the patient);
* Refer to the national standard for Clinic terminology of traditional Chinese medical diagnosis and treatment-Part 2:Syndromes/patterns, syndrome of "damp heat spleen" and "spleen deficiency with water stop" (Fulfill 2 of the main symptoms and 2 of the secondary symptoms).

Exclusion Criteria:

* Patients with a history of allergy to traditional Chinese medicine or Yunzhi;
* Patients who required nasal feeding or difficulty swallowing;
* Patients with comatose/semi-conscious, cognitively impaired with dementia/confusion, physically too ill with extremely poor general condition, or there was a language barrier.

Ages: 21 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Score change of McGilll QOL-Hong Kong | 6 months
  McGill QOL-Hong Kong questionnaire will be used to measure the quality of life of subjects. It consists of 16 items and also a single item rating the overall QOL. All the response categories are based on a numerical scale from 0 to 10, with verbal anchors at the ends of the scale. The higher the score, the better the quality of life.

SECONDARY OUTCOMES:
Survival rate | From baseline to 6 months
  Survival rate will be measured from baseline to month 6
Changes in immunological levels | 4 months
  T Serum immunoglobulins levels such as immunoglobulin A (IgA), immunoglobulin G (IgG) and immunoglobulin M (IgM) are key immunological markers for the humoral immune status. The levels of IgA, IgG and IgM are determined routinely in clinical practice to give the doctors important information about the immune system function, especially relating to infection or autoimmune diseases.
Changes in immunological levels | 6 months
  T Serum immunoglobulins levels such as immunoglobulin A (IgA), immunoglobulin G (IgG) and immunoglobulin M (IgM) are key immunological markers for the humoral immune status. The levels of IgA, IgG and IgM are determined routinely in clinical practice to give the doctors important information about the immune system function, especially relating to infection or autoimmune diseases.
Changes in tumor marker level | 4 months
  When cancer occurs, a substance called "tumor marker" will appear in the body. It may be a by-product of cancer cells or the body's response to the tumor. Most tumor markers are proteins that can be detected in blood or urine come out. Tumor markers help to determine the possibility of cancer in some patients. One of the most important uses of tumor markers is to monitor the progress of patients during treatment.
  The blood sample will be taken for measuring the tumor marker on month 4.
Changes in tumor marker level | 6 months
  When cancer occurs, a substance called "tumor marker" will appear in the body. It may be a by-product of cancer cells or the body's response to the tumor. Most tumor markers are proteins that can be detected in blood or urine come out. Tumor markers help to determine the possibility of cancer in some patients. One of the most important uses of tumor markers is to monitor the progress of patients during treatment.
  The blood sample will be taken for measuring the tumor marker on month 6.
Score change of Edmonton Symptom Assessment System (ESAS) | 6 months
  The ESAS includes 11 common patient symptoms: pain, tiredness, nausea, depression, anxiety, drowsiness, appetite, sleep, well-being, shortness of breath, and "other". It uses a 0-10 numerical scale: 0 indicates the absence of a symptom, and 10 indicates the worst experience of the symptom.
Use of rescue pain medication | From baseline to 6 months
  Number of rescue pain medication will be record during the study period
Number of interventional medical treatments | From baseline to 6 months
  Total number of interventional medical treatment will be records during the study period
Level change of total bilirubin | From baseline to 6 months
  Blood samples will be taken for Liver function test(LFT). Total bilirubin will be measured.
Level change of Alkaline Phosphatase (ALP) | From baseline to 6 months
  Blood samples will be taken for Liver function test(LFT). Alkaline Phosphatase (ALP) will be measured.
Level change of Alanine Transaminase (ALT) | From baseline to 6 months
  Blood samples will be taken for Liver function test(LFT). Alanine Transaminase (ALT) will be measured.
Level change of Aspartate Transferase (AST) | From baseline to 6 months
  Blood samples will be taken for Liver function test(LFT). Aspartate Transferase (AST) will be measured.
Level change of Gamma-glutamyl Transferase (GGT) | From baseline to 6 months
  Blood samples will be taken for Liver function test(LFT). Gamma-glutamyl Transferase (GGT) will be measured.
Level change of Creatinine | From baseline to 6 months
  Blood samples will be taken for Renal function test (RFT). Creatinine will be measured.
Level change of Sodium | From baseline to 6 months
  Blood samples will be taken for Renal function test (RFT). Sodium will be measured.
Level change of Potassium | From baseline to 6 months
  Blood samples will be taken for Renal function test (RFT). Potassium will be measured.
Level change of Blood urea nitrogen (BUN) | From baseline to 6 months
  Blood samples will be taken for Renal function test (RFT). Blood urea nitrogen (BUN) will be measured.
Level change of Uric acid | From baseline to 6 months
  Blood samples will be taken for Renal function test (RFT). Uric acid will be measured.
Level change of blood markers | From baseline to 6 months
  Blood samples will be taken for Complete blood count (CBC)
Change of urine analysis | 2 months
  Urine sample will be taken for urine protein analysis.
Change of urine analysis | 4 months
  Urine sample will be taken for urine protein analysis.
Change of urine analysis | 6 months
  Urine sample will be taken for urine protein analysis.
Change in body weight | From baseline to 6 months
  Body weight will be measure during each visit
Number of oral ulcer | From baseline to 6 months
  Total number of oral ulcer during study period
Change in Chinese medicine symptom score | 2 months
  Chinese medicine practitioners will assess subjects' symptoms in month 2, the symptoms such as bloating, less appetite, fatigue and defecation.
  The symptoms will be scored on a scale of 0,2,4,6, which represents none, mild, moderate and severe respectively. A higher score means a worse outcome.
Change in Chinese medicine symptom score | 4 months
  Chinese medicine practitioners will assess subjects' symptoms in month 4, the symptoms such as bloating, less appetite, fatigue and defecation.
  The symptoms will be scored on a scale of 0,2,4,6, which represents none, mild, moderate and severe respectively. A higher score means a worse outcome.
Change in Chinese medicine symptom score | 6 months
  Chinese medicine practitioners will assess subjects' symptoms in month 6, the symptoms such as bloating, less appetite, fatigue and defecation.
  The symptoms will be scored on a scale of 0,2,4,6, which represents none, mild, moderate and severe respectively. A higher score means a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Zhixiu Lin, Principal Investigator — Hong Kong Institute of Integrative Medicine